CLINICAL TRIAL: NCT06385600
Title: Intravenous Labetalol Versus Phentolamine for the Management of Severe Preeclampsia , Randomized Controlled Clinical Trial
Brief Title: Intravenous Labetalol vs Phentolamine for the Management of Severe Preeclampsia.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Mostafa, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: severe preeclampsia
Record Dates: First submitted 2024-02-08; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Severe Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Labetalol; halofantrine; Phentolamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- labetalol in the managment of severe preeclampsia (Active Comparator): labetalol intravenous infusion (Trandate, Gsk) in a concentration of 10 mg/ ml, thus 50 mg/ml equals to 5 ml/hr. The starting infusion rate of the antihypertensive medication is 5 ml/hr for an 80 Kg patient
  Interventions: Drug: Labetalol
- phentolamine in the managment of severe preeclampsia (Active Comparator): phentolamine intravenous infusion (Rogitamine) in a concentration of 10 mg/ml, thus 1 µg/Kg/min equals to 4.8 ml/hr for an 80 Kg patient
  Interventions: Drug: Phentolamine

INTERVENTIONS:
Drug: Labetalol — Group L will recieve labetalol intravenous infusion (Trandate, Gsk) in a concentration of 10 mg/ ml, thus 50 mg/ml equals to 5 ml/hr. The starting infusion rate of the antihypertensive medication is 5 ml/hr for an 80 Kg patient.
  Other Names: trandate, Gsk
  Arms: labetalol in the managment of severe preeclampsia
Drug: Phentolamine — Group P will receive phentolamine intravenous infusion (Rogitamine) in a concentration of 10 mg/ml, thus 1 µg/Kg/min equals to 4.8 ml/hr for an 80 Kg patient.
  Other Names: Rogitamine
  Arms: phentolamine in the managment of severe preeclampsia

SUMMARY:
The only effective treatment of severe preeclampsia is delivery of the fetus but immediate antihypertensive treatment is given to stabilize the patient and prevent further complications. All antihypertensive medication can potentially cross the placenta. At this time, there are no randomized control trials to base a recommendation for the use of one antihypertensive agent over another. However, certain medications are effective in lowering blood pressure with an acceptable safety profile in pregnancy. The choice of therapy depends on the acuity and severity of hypertension

DETAILED DESCRIPTION:
Non-invasive assessment of cerebral haemodynamics using Transcranial doppler ultrasonography has recently gained importance. Essentially, TCD measures flow velocity in the insonated vessel and the changes in flow velocity can be taken to reflect the changes in blood flow, assuming that the diameter of the insonated vessel remains constant. As TCD is easy to use and gives reproducible measurements, it has become a widely accepted method of assessing the cerebrovascular reactivity to carbon dioxide (CRCO2), cerebral autoregulation, estimated CPP, and CrCP. In patients with neurological disorders, impairment in both cerebral autoregulation and cerebral vascular reactivity has been shown to predict poor neurological outcome. Knowledge of the effects of normal pregnancy and pre-eclampsia on cerebral haemodynamics is essential for appropriate management of these patients undergoing anaesthesia or in labour, particularly when vasoactive medications are administered. The effects of pregnancy and/or pre-eclampsia on MCAFV have been studied by other investigators. Ikeda and colleagues found little change in mean MCAFV during the first two trimesters but reduced values in the third trimester. Williams and Wilson showed that MCAFV fell significantly with advancing gestational age. In another study, Williams and Wilson used TCD to assess cerebral haemodynamics in 17 non-pregnant women, 17 normotensive pregnant women, 20 pregnant women with pre-existing hypertension, and 21 pre-eclamptic women. The pregnant women were all in their third trimester. There was no difference in mean MCAFV in healthy pregnancy compared with non-pregnant women and a small, but non-significant, increase in mean MCAFV in the hypertensive and pre-eclamptic women. Demarin and colleagues studied pre-eclamptic women before and after delivery and found a progressive increase in MCAFV during late pregnancy. Ohno and colleagues compared MCAFV in 35 healthy pregnant and 17 pre-eclamptic women. In this study, the mean MCAFV was significantly higher in the pre-eclamptic group. It has been suggested that these increases in MCAFV are because of a degree of vasospasm. The differences between the findings of various studies with regards to the changes in MCAFV in pre-eclampsia might be explained by the differences in the severity of pre-eclampsia between the studies. Some investigators have reported increased MCAFV in symptomatic, compared with asymptomatic pre-eclamptics.

ELIGIBILITY:
Inclusion Criteria:

* • Pregnant woman with severe preeclampsia diagnosed by obstetric doctor

  * Patients willing to participate in the study
  * Age above 18 yrs

Exclusion Criteria:

* • Patients with eminent eclampsia

  * The history of optic neuritis
  * Severe myopia
  * History of ocular surgeries
  * Presence of ocular ulcers
  * Any clinical or morphological conditions that prevent the ultrasound examination of the orbital area
  * Age below 18 yrs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
the effect of Labetalol and Phentolamine on MCA flow velocity by transcranial Doppler monitoring. | 6 hours
  Singleton pregnant women who suffered from late onset preeclampsia will be enrolled and subjected to baseline Transcranial doppler (TCD) evaluation to measure middle cerebral artery (MCA) blood flow indices including mean flow velocity (cm/s).

SECONDARY OUTCOMES:
The effect of labetalol and phentolamine on blood pressure of the patients | 6 hours
  through measuring the blood pressure in (mmHg)